CLINICAL TRIAL: NCT01403142
Title: Optical Coherence Tomography to Evaluate Cardiac Allograft Vasculopathy in Patients Undergoing Clinically Indicated Angiographies Post Heart Transplant
Brief Title: Optical Coherence Tomography (OCT) to Evaluate Cardiac Allograft Vasculopathy (CAV) in Patient's Post Heart Transplant
Acronym: OCTCAV
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Tamim Nazif, Assistant Professor of Medicine, Columbia University
Other Study IDs: AAAI1023
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: heart transplant; vasculopathy
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac allograft vasculopathy (CAV) is a unique form of accelerated plaque formation seen in the coronary arteries of patients who have received heart transplantation. It is a major cause of morbidity and mortality in patients after heart transplant. Little progress has been made in characterizing this disease process, with more sophisticated imaging allowing for more detailed analysis of CAV, superior stratification of transplant recipients is possible and earlier interventions can be performed if necessary to prevent mortality and graft loss.

Optical Coherence Tomography (OCT) is a novel imaging modality with much higher resolution then Intra-Vascular Ultrasound (IVUS). This study will involve examining patients post-heart transplant using this high-resolution imaging modality. It is currently the standard care for patients post-heart transplant to receive annual coronary angiograms with close follow up. Patients will be imaged using OCT at the time of their routine annual angiogram, and will be re-imaged one year later at the time of the next annual angiogram or earlier if clinically indicated. The study goal is to better characterize CAV in vivo with OCT imaging and to try to identify patterns of the disease, including intra-coronary risk assessment.

DETAILED DESCRIPTION:
This study will involve imaging up to 100 patients at different points in time post heart transplant as part of their standard of care, with various degrees of disease and with different lesion subtypes. Imaging will take place at the time of routine coronary angiogram, which is standard of care in this patient population,or when clinically indicated. In prior studies using IVUS todetect CAV, the yield was significantly higher with multi-vessels imaged. OCT is an intravascular light-based imaging modality that measures the intensity of reflected light waves and converts these echoes into a high-resolution tomographic image. It is a catheter-based invasive imaging system analogous to IVUS but uses light as opposed to ultrasound to generate in vivo images of coronary arteries. It has the highest resolution of any intravascular imaging modality, capable of obtaining detailed cross-sectional images of coronary arteries in vivo at a resolution of 10 um or near histologic. This device, which is FDA approved for intracoronary evaluation, has been used in evaluating patients with coronary artery disease, specifically for plaque composition analysis, as well as for proper stent deployment after percutaneous intervention.

ELIGIBILITY:
Inclusion Criteria:

* Post heart transplant patients
* Patients presenting for their routine annual or clinically indicated coronary angiogram post-heart transplant. The decision for coronary angiogram will be made by the treating physician from the heart-failure-transplant team (not by the physician who will do the angiogram)
* Clinically suspect or evidence of CAV in previous coronary angiogram
* Age > 18
* Written informed-consent obtained

Exclusion Criteria:

* Any complications that occur during routine biopsy of the coronary arteries during the same cath-lab visit
* Baseline renal failure with Cr > 1.8
* Contraindication for anticoagulation
* Any other condition that in the opinion of the investigators would alter the safety of participation, or interfere with the ability to adhere to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-08-18 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Oberservational study. There are no specific outcome measures | prior to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Nazif, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong L, Maehara A, Nazif TM, Pollack AT, Saito S, Rabbani LE, Apfelbaum MA, Dalton K, Moses JW, Jorde UP, Xu K, Mintz GS, Mancini DM, Weisz G. Optical coherence tomographic evaluation of transplant coronary artery vasculopathy with correlation to cellular rejection. Circ Cardiovasc Interv. 2014 Apr;7(2):199-206. doi: 10.1161/CIRCINTERVENTIONS.113.000949. Epub 2014 Apr 8. PMID 24714488